CLINICAL TRIAL: NCT03162653
Title: Effect of ALlopurinol in Addition to Hypothermia for Hypoxic-ischemic Brain Injury on Neurocognitive Outcome - a Blinded Randomized Placebo-controlled Parallel Group Multicenter Trial for Superiority (Phase III)
Brief Title: Effect of Allopurinol for Hypoxic-ischemic Brain Injury on Neurocognitive Outcome
Acronym: ALBINO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Technische Universität Dresden (Other); UMC Utrecht (Other); KU Leuven (Other); University of Zurich (Other); University of Vienna (Other); Fundación para la Investigación del Hospital Clínico de Valencia (Other); Universidade do Porto (Other); Oslo University Hospital (Other); Università degli Studi di Udine (Unknown); Helsingin Ja Uudenmaan Sairaanhoitopiirin (Unknown); University of Helsinki (Other); Poznan University of Medical Sciences (Other); Tartu University Hospital (Other); ACE Pharmaceuticals BV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALBINO; 2016-000222-19 (EudraCT Number)
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Encephalopathy, Hypoxic-Ischemic; Infant, Newborn, Diseases
Keywords: Allopurinol; hypothermia therapy; hypoxic-ischemic encephalopathy; neonatal oxygen deficiency; childbirth outcome; perinatal asphyxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Infant, Newborn, Diseases | interventions — Allopurinol; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allopurinol (Active Comparator): Allopurinol, powder for injection (PFI), administered in two doses. First dose (20 mg/kg in 2ml/kg sterile water for injection) given as soon as intravenous access is established and no later than 30min postnatally and second dose (10mg/kg in 1ml/kg sterile water for injection) 12 hours thereafter. The second dose will only be administered to in infants on therapeutic hypothermia. Infants who recover quickly and do not qualify for and hence do not undergo hypothermia will not receive a second dose. Administration will be by continuous infusion using a syringe pump over 10min through secure venous access.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): mannitol, powder for injection (PFI), administered in two doses. First dose (20 mg/kg in 2ml/kg sterile water for injection) given as soon as intravenous access is established and no later than 30min postnatally and second dose (10mg/kg in 1ml/kg sterile water for injection) 12 hours thereafter. The second dose will only be administered to in infants on therapeutic hypothermia. Infants who recover quickly and do not qualify for and hence do not undergo hypothermia will not receive a second dose. Administration will be by continuous infusion using a syringe pump over 10min through secure venous access.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol, powder for injection (PFI), administered in two doses. First dose (20 mg/kg in 2ml/kg sterile water for injection) given as soon as intravenous access is established and no later than 30min postnatally and second dose (10mg/kg in 1ml/kg sterile water for injection) 12 hours thereafter. The second dose will only be administered to in infants on therapeutic hypothermia. Infants who recover quickly and do not qualify for and hence do not undergo hypothermia will not receive a second dose. Administration will be by continuous infusion using a syringe pump over 10min through secure venous access.
  Arms: Allopurinol
Drug: Mannitol — Placebo (Mannitol, PFI, 20mg/kg in the same volume and at the same time intervals as the intervention group - (2nd dose 10mg/kg only if infant undergoes therapeutic hypothermia)).
  Arms: Placebo

SUMMARY:
Neonatal hypoxic-ischemic encephalopathy (HIE) is a major cause of death or long-term disability in infants born at term in the western world, affecting about 1-4 per 1.000 life births and consequently about 5-20.000 infants per year in Europe.

Hypothermic treatment became the only established therapy to improve outcome after perinatal hypoxic-ischemic insults. Despite hypothermia and neonatal intensive care, 45-50% of affected children die or suffer from long-term neurodevelopmental impairment. Additional neuroprotective interventions, beside hypothermia, are warranted to further improve their outcome.

Allopurinol is a xanthine oxidase inhibitor and reduces the production of oxygen radicals and brain damage in experimental, animal, and early human studies of ischemia and reperfusion.

This project aims to evaluate the efficacy and safety of allopurinol administered immediately after birth to near-term infants with HIE in addition to hypothermic treatment.

DETAILED DESCRIPTION:
During labour and childbirth various events (such as placental abruption, uterine rupture, umbilical cord complications etc.) may result in impaired oxygenation and/or perfusion of the newborn brain which may result in brain injury termed "hypoxic-ischemic encephalopathy" (HIE). HIE is associated with development of long-term motor, cognitive, and neurosensory and memory disability and is one of the fundamental problems in perinatal medicine affecting about 5,000-20,000 infants/year in Europe (or 1-4/1000 live births in western societies) and approximately 1 million infants/year worldwide.

In term infants with perinatal asphyxia and postnatal HIE, brain injury predominantly originates in the immediate perinatal period (in contrast to a more distant prenatally acquired brain injury) as indicated by the lack of already established brain injury on early postnatal MRI. Consequently, brain injury in this population may potentially be ameliorated by postnatal pharmacological interventions.

The most common motor disability resulting from HIE is "cerebral palsy", the other major adverse outcome is cognitive disability, which prevents affected patients to lead their lives independently (without assistance and/or financial support).

The single major cause of HIE is a perinatal hypoxic/ischemic event (perinatal asphyxia). This hypoxic insult can cause immediate (necrosis) and delayed death (apoptosis) of (especially neuronal) cells, the latter responsible for a substantial amount of HIE-associated permanent brain damage. Whereas no intervention is known to prevent necrosis, the delayed cell death by apoptosis can be reduced by therapeutic interventions: Apoptosis is in part caused by secondary energy failure which can be reduced by hypothermic treatment.

Apoptosis is also caused by xanthine oxidase-mediated production of cytotoxic oxygen radicals during reperfusion, and there is evidence that allopurinol, a xanthine-oxidase inhibitor, reduces delayed cell death in animal models of perinatal asphyxia and ischemia/reperfusion.

Allopurinol prevents adenosine degradation, oxygen radical formation, preserves NMDA receptor integrity, and consequently may reduce brain injury in HIE by several mechanisms of action which are independent from the proven beneficial effect of hypothermic treatment on cellular energy metabolism. An additional beneficial (or even synergistic?) effect of allopurinol in addition to hypothermia can therefore be expected.

As no safety concerns were known at the start of this study regarding administration of even high doses of Allopurinol to neonates a phase III study was planned instead of a pilot study or an adaptive design. Close follow-up of MR-imaging along with reporting of all safety relevant data to a Data Monitoring Committee (which includes experts for brain imaging not otherwise involved in the study) ensures patients' safety.

Primary objective of this study is to evaluate whether newborns with asphyxia and early clinical signs of hypoxic ischemic encephalopathy will benefit from early administered Allopurinol compared to placebo, both in addition to standard of care, regarding long-term follow-up such as severe neurodevelopmental impairment or death at two years.

ELIGIBILITY:
Inclusion criteria

Term and near-term infants with a history of disturbed labour who meet at least one criterion of perinatal acidosis (or ongoing resuscitation) and at least two early clinical signs of potentially evolving encephalopathy as defined herein:

Severe perinatal metabolic acidosis or ongoing cardiopulmonary resuscitation at 5 min after birth:

At least 1 out of the following 5 criteria must be met

* Umbilical (or arterial or reliable venous) blood gas within 30 min after birth with pH<7.0
* Umbilical (or arterial or reliable venous) blood gas within 30 min after birth with base deficit ≥16 mmol/l
* Need for ongoing cardiac massage at/beyond 5 min postnatally
* Need for adrenalin administration during resuscitation
* APGAR score ≤5 at 10min AND

Early clinical signs of potentially evolving encephalopathy:

At least 2 out of the following 4 criteria must be met:

* Altered state of consciousness (reduced or absent response to stimulation or hyperexcitability)
* Severe muscular hypotonia or hypertonia,
* Absent or insufficient spontaneous respiration (e.g., gasping only) with need for respiratory support at 10 min postnatally
* Abnormal primitive reflexes (absent suck or gag or corneal or Moro reflex) or abnormal movements (e.g., potential clinical correlates of seizure activity)

Exclusion criteria

* gestational age below 36 weeks
* birth weight below 2500 g
* postnatal age >30min at the end of screening phase
* severe congenital malformation or syndrome requiring neonatal surgery or affecting long-term outcome
* patient considered "moribund" / "non-viable" (e.g., lack of spontaneous cardiac activity and ongoing chest compression at 30min)
* decision for "comfort care only" before study drug administration
* parents declined study participation as response to measures of community engagement
* both parents are insufficiently fluent in the study site's national language(s) or English or do not seem to have the intellectual capacity to understand the study procedures and to give consent as judged by the personnel who had been in contact with the mother/father before delivery.
* both parents/guardians less than 18 years of age, in case of single parent/guardian this one less than 18 years of age

Max Age: 45 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 760 (Estimated)
Dates: Start 2018-03-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
death versus severe neurodevelopmental impairment versus survival without severe neurodevelopmental impairment | at the age of 24 months
  Where severe neurodevelopmental impairment is defined as any of the following: cognitive or language delay defined as a cognitive-composite-score or a language-composite-score on the Bayley Scales of Infant and Toddler Development (3rd edition) < 85 and/or cerebral palsy (CP) according to SCPE criteria [SCPE Dev Med Child Neurol 2000]. In case of missing Bayley III test results, Bayley II or other developmental test results or PARCA-R parent questionnaire results may substitute for the Bayley III test result in a predefined hierarchical order.
  Primary endpoint with three mutually exclusive responses (healthy, death, composite outcome for impairment) will be analyzed in the two treatment groups by a generalized logits model according to Bishop, Fienberg, Holland 1975 with SAS 9.4 procedure proc catmod.

SECONDARY OUTCOMES:
Death or neurodevelopmental impairment (NDI) | at 24months
  The primary endpoint will be reconstituted as dichotomised composite secondary endpoint (survival without NDI versus Death or language-composite-score < 85 or cognitive-composite score <85 or cerebral palsy present). In case of missing Bayley III test results, Bayley II or other developmental test results or PARCA-R parent questionnaire results may substitute for the Bayley III test result in a predefined hierarchical order.
  This will be analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Incidence of Death | at 24 months
  Incidence of death will be analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Incidence of CP | at 24 months
  Incidence of CP according to SCPE criteria [SCPE Dev Med Child Neurol 2000] will be analyzed by Cochrane-Mantel-Haenszel- X²-Test.
GMFCS-score | at 24 months
  GMFCS-Score for quantification of the effects of cerebral palsy and other motor impairments (adapted from Palisano et al. [Palisano Med Child Neurol 1997]) using the ALBINO-GMFCS-score sheet will be analysed. GMFCS-score consists of six categories. Analysis will be done by using Wilcoxon-Mann-Whitney test.
Motor-Composite-Score (Bayley III) | at 24 months
  The numerical data of the motor-composite-score will be analysed using Wilcoxon-Mann-Whitney test. The use of this test accounts for the fact that data will be cut due to lack of sensitivity below 50 points.
Motor-Composite-Score dichotomised (Bayley III) | at 24 months
  The motor-composite-score will be dichotomised at the cut-off <85 versus ≥85 and analysed by Cochrane-Mantel-Haenszel- X²-Test.
Cognitive-Composite-Score (cognitive subscale, Bayley III) | at 24 months
  The numerical data of the cognitive-composite-score will be analysed using Wilcoxon-Mann-Whitney test. The use of this test accounts for the fact that data will be cut due to lack of sensitivity below 50 points.
Cognitive-Composite-Score dichotomised (cognitive subscale, Bayley III) | at 24 months
  The cognitive-composite-score will be dichotomised at the cut-off <85 versus ≥85 and analysed by Cochrane-Mantel-Haenszel- X²-Test.
Language-Composite-Score (language subscale, Bayley III) | at 24 months
  The raw numerical data of the language-composite-score will be analysed using Wilcoxon Mann-Whitney test. The use of this test accounts for the fact that data will be cut due to lack of sensitivity below 50 points.
Language-Composite-Score dichotomised (language subscale, Bayley III) | at 24 months
  The language-composite-score will be dichotomised at the cut-off <85 versus ≥85 and analysed by Cochrane-Mantel-Haenszel- X²-Test

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, Prof. Dr., Study Director — University Children's Hospital Tuebingen; Rüdiger Mario, Prof. Dr., Principal Investigator — University Children's Hospital Dresden
Locations (12):
- Medizinische Universitaet Wien, Vienna, Austria
- Katholieke Universiteit Leuven, Leuven, Belgium
- Tartu Ulikool, Tartu, Estonia
- Helsingin Ja Uudenmaan Sairaanhoitopiirin Kuntayhtymä, Helsinki, Finland
- University Hospital Tübingen, Tübingen, Germany
- Universita Degli Studi Di Udine, Udine, Italy
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Oslo Universitetssykehus Hf, Oslo, Norway
- Uniwersytet Medyczny Im Karola Marcinkowskiego W Poznaniu, Poznan, Poland
- Universidade Do Porto, Porto, Portugal
- Para La Investigacion Del Hospital UniversitarioLa Fe De La Comunidad Valenciana, Valencia, Spain
- Universitaet Zuerich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maiwald CA, Annink KV, Rudiger M, Benders MJNL, van Bel F, Allegaert K, Naulaers G, Bassler D, Klebermass-Schrehof K, Vento M, Guimaraes H, Stiris T, Cattarossi L, Metsaranta M, Vanhatalo S, Mazela J, Metsvaht T, Jacobs Y, Franz AR; ALBINO Study Group. Effect of allopurinol in addition to hypothermia treatment in neonates for hypoxic-ischemic brain injury on neurocognitive outcome (ALBINO): study protocol of a blinded randomized placebo-controlled parallel group multicenter trial for superiority (phase III). BMC Pediatr. 2019 Jun 27;19(1):210. doi: 10.1186/s12887-019-1566-8. PMID 31248390
- [Background] Annink KV, Franz AR, Derks JB, Rudiger M, Bel FV, Benders MJNL. Allopurinol: Old Drug, New Indication in Neonates? Curr Pharm Des. 2017;23(38):5935-5942. doi: 10.2174/1381612823666170918123307. PMID 28925896
- [Background] Deferm N, Annink KV, Faelens R, Schroth M, Maiwald CA, Bakkali LE, van Bel F, Benders MJNL, van Weissenbruch MM, Hagen A, Smits A, Annaert P, Franz AR, Allegaert K; ALBINO Study Group. Glomerular Filtration Rate in Asphyxiated Neonates Under Therapeutic Whole-Body Hypothermia, Quantified by Mannitol Clearance. Clin Pharmacokinet. 2021 Jul;60(7):897-906. doi: 10.1007/s40262-021-00991-6. Epub 2021 Feb 21. PMID 33611729
- [Derived] Engel C, Rudiger M, Benders MJNL, van Bel F, Allegaert K, Naulaers G, Bassler D, Klebermass-Schrehof K, Vento M, Vilan A, Falck M, Mauro I, Metsaranta M, Vanhatalo S, Mazela J, Metsvaht T, van der Vlught R, Franz AR; ALBINO Study Group. Detailed statistical analysis plan for ALBINO: effect of Allopurinol in addition to hypothermia for hypoxic-ischemic Brain Injury on Neurocognitive Outcome - a blinded randomized placebo-controlled parallel group multicenter trial for superiority (phase III). Trials. 2024 Jan 24;25(1):81. doi: 10.1186/s13063-023-07828-6. PMID 38267942
- See also: official study homepage — http://www.albino-study.eu